CLINICAL TRIAL: NCT06568289
Title: Lignocaine vs Bupivacaine Infiltration for Postpartum Perineal Pain After Vaginal Delivery With Episiotomy in Primigravidae: A Prospective Randomized, Double-Blind, Clinical Trial
Brief Title: Lignocaine vs Bupivacaine Infiltration for Postpartum Perineal Pain After Vaginal Delivery With Episiotomy in Primigravidae
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mostafa Serry, Captain Doctor, Resident of Obstetrics and Gynecology-The Police academy hospitals, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMASUMS167/2024
Record Dates: First submitted 2024-08-21; First posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Lignocaine; Bupivacaine; Postpartum Perineal Pain; Vaginal Delivery; Episiotomy; Primigravidae
MeSH Terms: interventions — Lidocaine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lignocaine group (Experimental): A perineal infiltration of a 5-ml of the drug (100 mg of lignocaine) in the margins of the episiotomy. Careful aspiration before and during injection of the product should be performed to prevent intravascular injection. The entire contents will then be injected slowly at several points of infiltration. All planes will be infiltrated (vagina, muscle, and skin) before episiotomy repair.
  Interventions: Drug: Lignocaine
- Bupivacaine group (Experimental): A perineal infiltration of a 5-ml of the study drug (20 mg of Bupivacaine) in the margins of the episiotomy. Careful aspiration before and during injection of the product should be performed to prevent intravascular injection. The entire contents will then be injected slowly at several points of infiltration. All planes will be infiltrated (vagina, muscle, and skin) before episiotomy repair.
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Lignocaine — A perineal infiltration of a 5-ml of the drug (100 mg of lignocaine) in the margins of the episiotomy. Careful aspiration before and during injection of the product should be performed to prevent intravascular injection. The entire contents will then be injected slowly at several points of infiltration. All planes will be infiltrated (vagina, muscle, and skin) before episiotomy repair.
  Arms: Lignocaine group
Drug: Bupivacaine — A perineal infiltration of a 5-ml of the study drug (20 mg of Bupivacaine) in the margins of the episiotomy. Careful aspiration before and during injection of the product should be performed to prevent intravascular injection. The entire contents will then be injected slowly at several points of infiltration. All planes will be infiltrated (vagina, muscle, and skin) before episiotomy repair.
  Arms: Bupivacaine group

SUMMARY:
In this study, we will compare the effect and safety of lignocaine versus bupivacaine infiltration for postpartum perineal pain after vaginal delivery with episiotomy in primigravidae.

DETAILED DESCRIPTION:
Episiotomy is the most common procedure used for dilatation of the vaginal opening for giving birth. Although episiotomy is associated with benefits for the mother, it may lead to short term and long-term disabilities, including postpartum perineal pain that is secondary to perineal tearing. The perineal pain experienced due to receiving an episiotomy is severe during the first few days after delivery, and it can lead to limitations in movement and difficulties with urination and defecation.

Bupivacaine is a long-acting local anesthetic that effectively reduces postoperative pain. In practice, bupivacaine is used for infiltration anesthesia, nerve blocks, epidural, and caudal anesthesia. It has a more selective effect on sensory nerve fibers as compared to motor nerve fibers, therefore is preferred in obstetrics.

Lignocaine infiltration, with the presence or absence of epidural anesthesia, is the most frequently employed local anesthetic in ameliorating postpartum perineal pain. It is a rapid-onset amide local anesthetic with a short duration of action lasting up to two hours.

ELIGIBILITY:
Inclusion Criteria:

* Primigravidae with the full term undergoing vaginal delivery with episiotomy.
* Pregnancies and singleton vertex cephalic fetuses.
* In the active phase of the first stage of labor.

Exclusion Criteria:

* Patients with history of drug allergies to study drugs as this will increase the risk of complications.
* Patients undergoing vaginal delivery under epidural or spinal anesthesia as they will affect post-operative pain and interfere with assessment of efficacy of local infiltration of the study drugs.
* Evidence of local infection at site of injection as this will interfere with the action of the study drug and will increase the risk of complications.
* Inability to cooperate as this will affect our assessment.
* Patient's refusal.
* Any intraoperative complications that will affect our outcome criteria (bleeding, organ injury) as they will affect patient's vital data and affect our assessment.
* Neurological comorbidities (chronic pain disorder, chronic systemic disease, neurological disorder, neuropathic pain) as they will need more analgesia.
* Drug abuse as they will be tolerant to the used analgesics.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Primigravidae women with the full term undergoing vaginal delivery with episiotomy.
Enrollment: 60 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Degree of pain | 6 hours postoperatively
  Degree of pain will be assessed using the visual analogue scale (VAS) is the scale that will be used to assess postoperative pain and its intensity. A respondent will select a whole number (0- 10 integers) that best reflects the intensity of her pain, 1-10 will be recorded.
  Postoperative analgesic effect will be assessed using numeric version of the visual analogue scale (VAS) after delivery and local anesthetic infiltration (immediately after delivery, after 2 hours, after 4 hours, and after 6 hours).

SECONDARY OUTCOMES:
The time till first analgesic requirement | 6 hours postoperatively
  The time till first analgesic (non-steroidal anti-inflammatory drugs (NSAIDs) requirement which is defined as the time (immediately after delivery, after 2 hours, after 4 hours and after 6 hours) after delivery and local anesthetic infiltration. Rescue analgesia of morphine will be given as 3 mg bolus if the visual analogue scale > 3 to be repeated after 30 min if pain persists until the visual analogue scale < 4. VAS will be assessed after delivery, after 2 hours, after 4 hours, and after 6 hours.
Total analgesics consumption | 12 hours postoperatively
  Total analgesics consumption over 12-hour period post-operative with mentioning the number and time of drugs given and the total dose of each drug post-operative (presented by hours post-operative).Rescue analgesia of morphine will be given as 3 mg bolus if the visual analogue scale > 3 to be repeated after 30 min if pain persists until the visual analogue scale < 4. VAS will be assessed after delivery, after 2 hours, after 4 hours, and after 6 hours.
Incidence of compilation | 6 hours postoperatively
  Incidence of compilation will be recorded such as as allergy, nausea, vomiting, fever, angioedema or respiratory distress.
Time of post-operative ambulation | 12 hours postoperatively
  Post-operative ambulation enhancement in the form of time of start of ambulation (in hours) starting from end of surgery- walking- climbing stairs will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.